CLINICAL TRIAL: NCT03960463
Title: Evaluation of Oxygen Delivery With TransCu O2 to Study Success Rate of Surgically Closed Wounds
Brief Title: EO2 Oxygen Delivery To Study Success Rate of Surgically Closed Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Electrochemical Oxygen Concepts, Inc. (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-41361
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Surgical Wound; Diabetes; Amputation Wound; Incision Wound; Peripheral Arterial Disease; Breast Cancer; Diabetic Foot
Keywords: Infection; Dehiscence; Necrotic tissue; Surgical Revision; Scar tissue; Wound Closure
MeSH Terms: conditions — Surgical Wound; Diabetes Mellitus; Peripheral Arterial Disease; Breast Neoplasms; Diabetic Foot; Infections; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): Participants will be provided with a Transcu O2 ® Oxygen delivery system at the surgical site for 4 weeks as supportive care.
  Interventions: Device: Transcu O2®
- Control (No Intervention): Participants will be placed in a standard dressing at the surgical site and will be followed for 4 weeks.

INTERVENTIONS:
Device: Transcu O2® — Participants randomized into study active group will be provided with a Transcu O2® at their surgical site and followed for 4 weeks.
  Arms: Active

SUMMARY:
The investigators will test the efficacy of the novel oxygen diffusion dressing allows delivery tissue oxygenation via TransCu O2® Oxygen Delivery System for use in caring for patients with surgically closed wounds.

The investigators hypothesize that using this novel oxygen diffusion dressing will reduce the likelihood of necrotic tissue as well as severe incisional scar post-surgical closure by improving transcutaneous oxygen levels during wound healing process. TransCu O2 Oxygen Delivery System is a novel wound healing therapy that promises to enhance tissue hydration, which in turn may lead to quick epithelialization essential to reduce the likelihood of formation of necrotic tissue and excessive scars.

DETAILED DESCRIPTION:
Surgical wound (e.g., post minor amputation, reconstruction surgery, or surgical incision) complications such as infection, dehiscence, necrotic tissue, surgical revision, and poor cosmesis are unfortunately highly prevalent in patients undergoing surgical interventions. In most cases surgical wounds are managed with a simple island dressing, orthopaedic wool padding and a light retention bandage. It could be argued that such low cost, traditional dressings are adequate for most surgical wounds. However, some patients with poor tissue integrity often require modern wound care products that offer additional benefits, in particular among those with vascular and poor tissue oxygenation problem. Poor tissue oxygenation and poor skin perfusion could lead to surgical wound complications such as wound infection, tissue necrosis, phantom pain, trauma and untimely surgical revision as well as major amputation.

In particular, the presence of non-viable, necrotic tissue (estimated to occur in 15-25% of cases) is significant as it can be responsible for delaying healing, prolonging the inflammatory response, mechanically obstructing contraction and impeding re-epithelialisation. It also provides a focus for wound infection and surgical revision.

The problem associated with necrotic tissue is not limited to limb amputation and could be seen in other surgical closures leading to excessive scar formation. Many of these scars can be problematic, being aesthetically unpleasant and causing discomfort. Blood supply is a significant factor in wound healing, and an area of the skin with rich supply of vasculature is known to heal to finer scars. Several studies have demonstrated that mild hypoxia (lack of transcutaneous oxygen) is present in early scars, moderate hypoxia in proliferative scars, and severe hypoxia in regressive scars. Oxygen levels then return to normal in mature scars, which is consistent along with the dynamic change in microvessel density. Therefore level of transcutaneous oxygen could be a determinant factor in formation of excessive scar formation.

Dressing materials are known to influence postoperative surgical wound healing and scar formation. A particular dressing that could promote wound hydration is key to ensure quick epithelialization and decrease excessive scar formation. The current standard of care in wound healing is to promote a moist wound environment by regular changing dressing and hydrate wound when needed. Some new advanced dressing and products have been also suggested with promising results in reducing excessive scar formation such as the use of silicone sheeting, hydrogel wound dressing, etc.

In this study, the investigators hypothesize that using novel oxygen diffusion dressing allows delivery tissue oxygenation via TransCu O2® Oxygen Delivery System will reduce the likelihood of necrotic tissue as well as severe incisional scar post-surgical closure by improving transcutaneous oxygen levels during wound healing process. TransCu O2 Oxygen Delivery System is a novel wound healing therapy that promises to enhance tissue hydration, which in turn may lead to quick epithelialization essential to reduce the likelihood of formation of necrotic tissue and excessive scars.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age. Ability to provide informed consent.
* Presence of a wound due to surgical intervention and closure.
* Subject or responsible caregiver is willing and able to maintain the required offloading (as applicable for the location of the wound) and applicable dressing changes

Exclusion Criteria:

* Charcot Arthropathy Bilateral AK/BK amputation Active Drug/alcohol abuse (or history of drug/alcohol abuse in last 1 month) Dementia or impaired cognitive function Subjects with osteomyelitis or extreme gangrene. Excessive lymphedema Presence of active infection Subject has a history of or any intercurrent illnesses or conditions that would compromise the safety of the subject according to judgement of a qualified wound specialist.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 22 | 11
Completed | 20 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 20 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We initially enrolled 33 participants (Active:22, Control:11). Two subjects in the active group withdrew consent after recruitment and prior to receiving the intervention. As a result, data from 20 participants in the active group were reported.
  years | 64.4 (10.6) | 64.6 (9.1) | 64.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We initially enrolled 33 participants (Active:22, Control:11). Two subjects in the active group withdrew consent after recruitment and prior to receiving the intervention. As a result, data from 20 participants in the active group were reported.
  Participants
    Female | 11 | 2 | 13
    Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We initially enrolled 33 participants (Active:22, Control:11). Two subjects in the active group withdrew consent after recruitment and prior to receiving the intervention. As a result, data from 20 participants in the active group were reported.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 7 | 3 | 10
    White | 8 | 6 | 14
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 11 | 31
CKD (Chronic Kidney Disease) [Count of Participants; unit: Participants] — Population: Diagnosis of CKD was unknown for two of participants out of 20
  Participants
    number analyzed (Participants) | 18 | 11 | 29
    (all) | 10 | 4 | 14
HbA1c [Mean (Standard Deviation); unit: % HbA1c] — Population: Two subjects in the active group withdrew consent after recruitment and prior to receiving the intervention. As a result, data from 20 participants in the active group were reported.
  % HbA1c | 9.4 (3.5) | 7.2 (.8) | 8.6 (3.0)
Type of Surgery [Count of Participants; unit: Participants] — Population: Two subjects in the active group withdrew consent after recruitment and prior to receiving the intervention. As a result, data from 20 participants in the active group were reported.
  Participants
    Toe amputations | 17 | 11 | 28
    Transmetatarsal amputation | 1 | 0 | 1
    Revision of amputation site | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unfavorable Wound Healing Outcomes at 4 Weeks
Description: Unfavorable wound healing outcomes were defined as the occurrence of one or more of the following conditions : infection, wound dehiscence, or necrotic tissue, as documented in the patient chart up to 4 weeks after the surgical wound closure.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 20 | 11
Participants | 8 | 7

2. Secondary Outcome: Length of Wound
Description: Length of surgical closed wound was measured using camera . The unit is cm
Time Frame: baseline and week 4
Population: Subjects with wound adhesive issues (e.g., wound re-opening) were excluded, and those with unavailable wound data at 4 weeks were not included
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Active | Control
Number analyzed (Participants) | 13 | 8
cm
  Baseline | 4.78 (3.36) | 4.28 (3.11)
  week 4 | 3.57 (2.92) | 7.28 (2.92)

3. Secondary Outcome: Change in Skin Perfusion at Baseline and 4 Weeks
Description: skin perfusion will be assessed Skin Perfusion Pressure Test (SPP)
Time Frame: baseline to 4 weeks
Population: The data for some participants were not available
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Active | Control
Number analyzed (Participants) | 14 | 11
mm Hg
  Baseline | 62.2 (18) | 72.3 (3.2)
  At 4 weeks | 63.1 (20) | 63.2 (19.9)

4. Secondary Outcome: Change in Percentage of Tissue Oxygen Saturation From Baseline to 4 Weeks
Description: Tissue oxygen saturation was assessed by a non-invasive tissue oxygenation measurement system (Snapshot, Kent Imaging)
Time Frame: baseline to 4 weeks
Population: Only participants with available data at baseline and 4 weeks were included
Measure: Mean (Standard Deviation); unit: Percentage of tissue oxygen saturation
Arm/Group | Active | Control
Number analyzed (Participants) | 14 | 11
Percentage of tissue oxygen saturation
  Baseline | 50 (19.9) | 56 (1.9)
  4 weeks | 50.6 (14.3) | 50 (21)

5. Secondary Outcome: Self-reported Pain at Week 4
Description: Pain will be assessed with visual analogue scale from 0 to 10 where 10 is the worst pain ever.
Time Frame: week 4
Population: Only participants with available data at week 4 were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 11 | 8
units on a scale | 2.09 (3.27) | 2.25 (1.98)

6. Secondary Outcome: Reintervention
Description: The need for podiatric reintervention (e.g., wound reclosure due to wound adhesive failure) within 30 days of surgical wound closure.
Time Frame: 4 weeks
Population: The data for one subject in the active group (out of the 20 subjects included) was unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 19 | 11
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: AEs were collected from study start date to the study completion date in a non-systematic way. Per patient, AEs were collected up to 4 weeks after baseline. During follow-ups, participants were asked if they experienced AEs. If participant missed a visit or had low adherence the coordinator called the participant and asked for AEs. AEs were also reported by the participants on a case-by-case basis when they occurred.
Description: The clinicaltrials.gov definitions were used. We collected unfavorable medical occurrences experienced by study participants and noted whether they were study device related (caused directly by the device), unrelated to the study device, or whether it was caused by improper device usage. This information was collected non-systematically and not separately -- either participants reported events directly or during phone calls/study visits study coordinators asked about issues.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/11
Other Adverse Events (participants affected / at risk) | 2/20 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=20) | Control (N=11)
Non-Study Related Adverse Event (General disorders) | 2 | 0 — 1 participant had their wound reopen after trauma to wound site (unrelated to study device) 1 participant had severe bleeding unrelated to study device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03960463/Prot_SAP_000.pdf